CLINICAL TRIAL: NCT00128219
Title: A Phase II Randomized, Double-Blinded, Comparative Clinical Trial for a Group B Streptococcus Serotype III-Tetanus Toxoid (GBS III-TT) Vaccine to Prevent Vaginal Acquisition of GBS Type III
Brief Title: Prevention of GBS Colonization Via Immunity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 02-015
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2009-08

CONDITIONS: Beta Haemolytic Streptococcal Infection
Keywords: Group B Streptococcus, women, vaccine
MeSH Terms: interventions — Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GBS III-TT (Experimental): A single dose of GBS III-TT vaccine administered intramuscularly (IM) containing 50 mcg of GBS III capsular polysaccharide and 32 mcg of tetanus toxoid.
  Interventions: Biological: GBS III-TT
- Td (Active Comparator): The control group will receive a single dose of Tetanus and Diphtheria Toxoids (Td) vaccine.
  Interventions: Biological: Tetanus and diptheria toxoids vaccine

INTERVENTIONS:
Biological: GBS III-TT — 50 mcg GBS Type III capsular polysaccharide conjugated to 32 mcg of tetanus toxoid. A single dose of vaccine administered by intramuscular (IM) injection in the upper arm. All subjects will receive a volume of 0.5 ml.
  Arms: GBS III-TT
Biological: Tetanus and diptheria toxoids vaccine — Td vaccine is a sterile solution of alum-precipitated toxoids in isotonic sodium chloride solution. A single dose of vaccine will be administered by intramuscular (IM) injection in the upper arm. All subjects will receive a volume of 0.5 ml. Each 0.5 ml dose is formulated to contain 5 Lf (flocculation units) of tetanus toxoid and 2 Lf of diphtheria toxoid.
  Arms: Td

SUMMARY:
The group B streptococcus (GBS) vaccine study is being done to see if a single vaccination with a GBS type III vaccine can stop women from getting GBS type III bacteria in the vagina. Approximately 600 women, ages 18-40, will be enrolled from the clinical sites participating in this study. Participants will be non-pregnant, sexually active (sex with a male at least once in the last 4 months), and GBS negative in the vagina or rectum at the screening visit. Participants will be randomly assigned to receive the experimental GBS type III vaccine or a licensed vaccine containing Tetanus and Diphtheria Toxoids (Td). Participants will be followed at one month, 2 months and every other month thereafter following vaccination (for vaginal and rectal swab collection and a blood draw) for 1½ years or a total of 10 post vaccination visits.

DETAILED DESCRIPTION:
Vaginal colonization is the single most important risk factor for transmission of group B Streptococcus (GBS) from mothers to neonates, resulting in neonatal sepsis and/or meningitis. The long-term goal of this study is to determine whether vaccine-induced serum antibody to type III GBS will be sufficient to prevent vaginal acquisition of type III GBS. This study is linked to Division of Microbiology and Infectious Diseases protocol 04-018. It is a randomized, double-blinded, comparative clinical trial among young (18-40 years old), non-pregnant, sexually active women who are not currently colonized vaginally or rectally with type III GBS, it will be conducted to evaluate the efficacy of a GBS type III-TT vaccine for prevention of type III GBS vaginal acquisition. The observation period for each patient will be 18 months following vaccination. The specific objectives are: enroll 600 women (previously screened within last 14 days in a GBS Screening Protocol) identified as GBS type III negative, vaginally and rectally; vaccinate 600 women randomized to a 1:1 ratio with 50 micrograms of type III GBS polysaccharide conjugated to tetanus toxoid (GBS III-TT) or licensed vaccine containing Tetanus and Diphtheria Toxoids adsorbed for adult use (Td); measure reactogenicity by subject report in a 7-day symptom diary and by 1-2 day follow-up telephone call; evaluate women at 1, 2, 4, 6, 8, 10, 12, 14, 16 and 18 months for serum antibody response. Blood will be obtained at each of these clinic follow-up visits and serum will be used to compare type III GBS specific antibody levels at baseline and follow-up; assess vaginal and rectal acquisition by GBS at months 1, 2, 4, 6, 8, 10, 12, 14, 16 and 18 months using specimens obtained at the clinic visits; compare women receiving GBS III-TT vaccine to women receiving Td vaccine with respect to the time to first vaginal culture positive for type III GBS; assess the relationship between person-level covariates, including features of the decrease of type III GBS antibody levels over time, and the time to first vaginal culture positive for type III GBS; and assess the effect of vaginal colonization by hydrogen peroxide (H2O2)-producing Lactobacillus, sexual activity, antibiotic usage, rectal colonization with GBS and demographic features as risk factors for acquisition of type III GBS, independent of serum antibody levels. The primary study endpoint will be the time to the first vaginal swab that is type III GBS culture positive, with all previous cultures negative for type III GBS, not just the immediately preceding culture. The secondary endpoints include: the proportion of vaginal swabs that are type III GBS culture positive; the proportion of subjects whose vaginal cultures are type III GBS culture negative throughout the study; the frequency of vaginal colonization with GBS serotypes Ia, Ib, II and V; the measurement of serum immunoglobulin (Ig)G antibody levels to type III GBS at 1, 2, 4, 6, 8, 10 12, 14, 16 and 18 months following vaccination; the measurement of post-vaccination antibody levels to type III GBS, stratified by pre-vaccination levels of native antibody; the frequency of local and systemic symptoms attributable to vaccination; and the density of type III GBS cultured from vaginal swabs at culture positive visits.

ELIGIBILITY:
Inclusion Criteria:

* Participated in and completed the group B Streptococcus (GBS) Screening Protocol
* Non-pregnant women
* Aged 18-40 years at time of the screening protocol
* Currently sexually active at time of enrollment (sex with a male at least once in the last 4 months)
* Current use of effective birth control methods and stated intention to use the method for at least the next 30 days
* Provision of written informed consent
* Intention to stay in the geographical area for the next 18 months
* Access to telephone

Exclusion Criteria:

* Group B Streptococcus (GBS) positive by culture (vaginal and/or rectal), or culture positive for streptococcal strains that cross-react with GBS typing sera (vaginal and/or rectal).
* Pregnancy (all women will receive a urine pregnancy prior to vaccination).
* Any condition which in the opinion of the investigator would pose a health risk to the subject or interfere with the evaluation of the vaccine.
* Serious underlying disease, which is known at the time of vaccination (including: immunodeficiency, active or chronic hepatitis, immunosuppressive conditions which require systemic steroid therapy, or treatment for a malignancy during the past year).
* Receipt of any vaccine, blood product, or experimental medicine within the past 30 days with the exception of a licensed inactivated influenza vaccine.
* Plans to receive any vaccine, blood product, or experimental medicine in the next 30 days with the exception of a licensed inactivated influenza vaccine.
* Use of any antimicrobial agent(s) (vaginal or systemic) for treatment of any condition within 7 days prior to study enrollment (including: Monistat, Gyne-Lotrimin, et cetera )
* History of hypersensitivity to tetanus toxoid vaccine.
* Tetanus toxoid immunization within the previous 12 months.
* Previous participation in a study in which participants received tetanus toxoid vaccine or vaccine against Group B Streptococcus.
* Spontaneous or surgical menopause.
* Nursing mother.
* Hypersensitivity to thimerosal.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 667 (Actual)
Dates: Start 2003-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Medical College of Georgia, Augusta, Georgia
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Planned Parenthood of Houston and Southeast Texas, Inc., Houston, Texas

REFERENCES:
- [Derived] Hillier SL, Ferrieri P, Edwards MS, Ewell M, Ferris D, Fine P, Carey V, Meyn L, Hoagland D, Kasper DL, Paoletti LC, Hill H, Baker CJ. A Phase 2, Randomized, Control Trial of Group B Streptococcus (GBS) Type III Capsular Polysaccharide-tetanus Toxoid (GBS III-TT) Vaccine to Prevent Vaginal Colonization With GBS III. Clin Infect Dis. 2019 May 30;68(12):2079-2086. doi: 10.1093/cid/ciy838. PMID 30281066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Young (ages 18 through 40), sexually active (sex at least once in the last 4 months), non-pregnant women from the surrounding communities and who were negative for vaginal and rectal colonization with type III group B streptococcus (GBS) were offered enrollment, between July 7, 2003 and August 8, 2006
Pre-assignment Details: Participants were screened for vaginal and rectal colonization with type III GBS and only those negative were offered enrollment
Groups:
- GBS III-TT Vaccine: The experimental arm received a single dose of vaccine administered intramuscularly (IM) containing 50 mcg of GBS III capsular polysaccharide and 32 mcg of tetanus toxoid (GBS III-TT).
- Td Vaccine: The control group received a single dose of tetanus and diptheria toxoids adsorbed for adult use (Td vaccine).
Period: Overall Study
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Started | 333 | 334
Completed | 264 | 263
Not Completed | 69 | 71

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GBS III-TT Vaccine | Td Vaccine | Total
Number analyzed (Participants) | 333 | 334 | 667
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 333 | 334 | 667
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.58) | 26.1 (5.68) | 26.2 (5.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 333 | 334 | 667
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 333 | 334 | 667

OUTCOME MEASURES:

1. Primary Outcome: The Time to First Vaginal Swab That is Type III GBS Culture Positive, With All Previous Cultures Negative for Type III GBS, Not Just the Immediately Preceding Culture.
Description: Time to first acquisition of vaginal type III GBS was calculated as time from vaccination to the mid-point of the interval of ascertainment, censored by either the end of the follow-up period, or the first of 2 or more consecutive missed visits. Vaginal type III GBS status at missed visits prior to censoring was imputed from the subsequent visit.
Time Frame: Time from vaccination to acquisition of vaginal type III GBS, up to 18 months post-vaccination.
Population: All enrolled participants with at least one post-enrollment efficacy assessment were included in the intention to treat (ITT) Efficacy Analysis Cohort. Women were included without regard to protocol adherence, and classified by treatment randomized rather than received.
Measure: Number; unit: Participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 325 | 325
Participants
  Month 0 to 2 at risk | 325 | 325
  Month 0 to 2 with GBS | 20 | 15
  Month 0 to 2 censored | 18 | 15
  Month 2 to 4 at risk | 287 | 295
  Month 2 to 4 with GBS | 5 | 6
  Month 2 to 4 censored | 13 | 7
  Month 4 to 6 at risk | 269 | 282
  Month 4 to 6 with GBS | 1 | 7
  Month 4 to 6 censored | 8 | 7
  Month 6 to 8 at risk | 260 | 268
  Month 6 to 8 with GBS | 3 | 8
  Month 6 to 8 censored | 10 | 9
  Month 8 to 10 at risk | 247 | 251
  Month 8 to 10 with GBS | 0 | 2
  Month 8 to 10 censored | 8 | 6
  Month 10 to 12 at risk | 239 | 243
  Month 10 to 12 with GBS | 0 | 7
  Month 10 to 12 censored | 4 | 12
  Month 12 to 14 at risk | 235 | 224
  Month 12 to 14 with GBS | 2 | 3
  Month 12 to 14 censored | 7 | 3
  Month 14 to 16 at risk | 226 | 218
  Month 14 to 16 with GBS | 2 | 3
  Month 14 to 16 censored | 4 | 3
  Month 16 to 18 at risk | 220 | 212
  Month 16 to 18 with GBS | 1 | 2
  Month 16 to 18 censored | 185 | 168
Statistical Analysis 1: Comparison: GBS III-TT Vaccine vs Td Vaccine; Time to first acquisition of vaginal type III GBS was analyzed by fitting a Cox Proportional Hazards model stratified by region to the data. The null hypothesis of no vaccine efficacy was tested by the stratified log-rank test (score test). The point and interval estimates for vaccine efficacy were obtained by transforming those for treatment effect in the model; Test type: Superiority or Other; p = 0.044, Regression, Cox — The a priori threshold for statistical significance was set at 0.05; The study was multi-center, and the Cox model was stratified by geographic region of the participating clinical sites; Vaccine Efficacy, VE=1-RR=1-exp(ß) = 36, 95% CI 2-sided [1 to 58] — Vaccine efficacy (VE) was defined as one minus the relative risk (RR), which was estimated by exponentiating the treatment parameter (ß) from the Cox model fit

2. Secondary Outcome: Geometric Mean Concentration (GMC) of Serum Immunoglobulin G (IgG) Antibody Levels to Type III GBS Post-Vaccination.
Description: The GMC was calculated from IgG antibody to type III GBS assay results on serum specimens obtained at clinic visits during the 18 month post-vaccination follow-up period. Results at missed visits prior to loss to follow-up/final visit were not imputed.
Time Frame: Prior to and at 1, 2, 4, 6, 8, 10, 12, 14, 16, and 18 months following vaccination.
Population: All enrolled participants with at least one post-enrollment efficacy assessment were included in the ITT Efficacy Analysis Cohort. Women were included without regard to protocol adherence, and classified by treatment randomized rather than received.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/ml
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 325 | 325
µg/ml
  Month 0 | 0.29 [0.25 to 0.35] | 0.31 [0.26 to 0.37]
  Month 1 | 12.35 [9.60 to 15.90] | 0.29 [0.24 to 0.35]
  Month 2 | 12.55 [9.95 to 15.81] | 0.30 [0.25 to 0.35]
  Month 4 | 9.58 [7.67 to 11.97] | 0.29 [0.24 to 0.34]
  Month 6 | 7.26 [5.84 to 9.03] | 0.29 [0.24 to 0.34]
  Month 8 | 6.63 [5.32 to 8.27] | 0.26 [0.22 to 0.32]
  Month 10 | 5.80 [4.64 to 7.24] | 0.28 [0.23 to 0.33]
  Month 12 | 5.16 [4.14 to 6.43] | 0.27 [0.22 to 0.32]
  Month 14 | 4.80 [3.84 to 6.00] | 0.26 [0.22 to 0.32]
  Month 16 | 4.57 [3.67 to 5.69] | 0.28 [0.23 to 0.34]
  Month 18 | 3.99 [3.22 to 4.94] | 0.27 [0.22 to 0.33]

3. Secondary Outcome: Number of Participants With Any Solicited Local and Systemic Symptoms.
Description: Participants maintained a diary card to report the occurrence of solicited local and systemic symptoms for 7 days after vaccination. Participants are counted if they indicated experiencing the symptom at any severity during the reporting period.
Time Frame: Safety surveillance during the 1st 7 days.
Population: The Safety Analysis Cohort is comprised of all vaccinated women, categorized according to the product received, regardless of their randomized assignment. Due to vaccination errors, the number of participants in the Td group for the Safety Analysis Cohort (n=337) exceeds the number randomized to this group (n=334).
Measure: Number; unit: Participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 326 | 337
Participants
  General Arm Pain | 175 | 223
  Local Redness | 27 | 40
  Local Swelling | 23 | 52
  Local Tenderness at Injection Site | 234 | 276
  Any Solicited Local Symptom | 251 | 294
  Chills | 30 | 33
  Headache | 130 | 118
  Elevated Oral Temperature (>37.4 degrees Celsius) | 33 | 32
  Malaise (Decreased energy) | 103 | 111
  Myalgia (General muscle aches) | 91 | 112
  Nausea | 55 | 61
  Any Solicited Systemic Symptom | 208 | 206
  Any Solicited Symptom | 282 | 307

4. Secondary Outcome: Mean Fold-Rise in Serum IgG Antibody Levels to Type III GBS Post-Vaccination
Description: Fold-rises compare the IgG antibody level at post-vaccination to that obtained just prior to vaccination, for each visit during the 18-month follow-up period. Assay results at missed visits prior to loss to follow-up/final visit were not imputed.
Time Frame: Prior to and at 1, 2, 4, 6, 8, 10, 12, 14, 16, and 18 months following vaccination.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 325 | 325
Ratio
  Month 0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Month 1 | 41.29 [34.70 to 49.12] | 0.99 [0.95 to 1.03]
  Month 2 | 41.06 [35.27 to 47.80] | 0.98 [0.94 to 1.02]
  Month 4 | 31.64 [27.35 to 36.60] | 0.93 [0.90 to 0.97]
  Month 6 | 25.56 [22.07 to 29.59] | 0.92 [0.88 to 0.97]
  Month 8 | 21.92 [18.95 to 25.36] | 0.89 [0.84 to 0.94]
  Month 10 | 19.78 [17.08 to 22.91] | 0.91 [0.87 to 0.96]
  Month 12 | 17.71 [15.30 to 20.50] | 0.91 [0.86 to 0.96]
  Month 14 | 16.76 [14.41 to 19.49] | 0.92 [0.87 to 0.98]
  Month 16 | 15.89 [13.70 to 18.42] | 0.90 [0.85 to 0.95]
  Month 18 | 14.26 [12.33 to 16.48] | 0.92 [0.87 to 0.97]

5. Secondary Outcome: Number of Participants With a Four-Fold or Greater Rise in Serum IgG Antibody to Type III GBS at Month 1 Post-Vaccination
Description: Blood samples were collected from participants prior to vaccination and at 1 month post vaccination, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The lower detection limit for the assay was 0.08 micrograms/milliliter (µg/mL), and antibody levels below this limit were recorded as 0.04 µg/mL by the laboratory. Fold rises compare IgG antibody levels at the post-vaccination visit to that obtained just prior to vaccination. Participants are considered a responder if the antibody increase was four-fold or greater.
Time Frame: Prior to and 1 month following vaccination
Population: All enrolled participants with blood collected at both time points were included in the ITT Efficacy Analysis Cohort. Women were included without regard to protocol adherence, and classified by treatment randomized rather than received.
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 304 | 303
participants | 277 | 1

6. Secondary Outcome: Number of Participants With a Four-Fold or Greater Rise in Serum IgG Antibody to Type III GBS at Month 2 Post-Vaccination
Description: Blood samples were collected from participants prior to vaccination and at 2 months post vaccination, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The lower detection limit for the assay was 0.08 micrograms/milliliter (µg/mL), and antibody levels below this limit were recorded as 0.04 µg/mL by the laboratory. Fold rises compare IgG antibody levels at the post-vaccination visit to that obtained just prior to vaccination. Participants are considered a responder if the antibody increase was four-fold or greater.
Time Frame: Prior to and 2 months following vaccination
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 301 | 310
participants | 286 | 1

7. Secondary Outcome: Number of Participants With a Four-Fold or Greater Rise in Serum IgG Antibody to Type III GBS at Month 4 Post-Vaccination
Description: Blood samples were collected from participants prior to vaccination and at 4 months post vaccination, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The lower detection limit for the assay was 0.08 micrograms/milliliter (µg/mL), and antibody levels below this limit were recorded as 0.04 µg/mL by the laboratory. Fold rises compare IgG antibody levels at the post-vaccination visit to that obtained just prior to vaccination. Participants are considered a responder if the antibody increase was four-fold or greater.
Time Frame: Prior to and 4 months following vaccination
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 289 | 298
participants | 272 | 2

8. Secondary Outcome: Number of Participants With a Four-Fold or Greater Rise in Serum IgG Antibody to Type III GBS at Month 6 Post-Vaccination
Description: Blood samples were collected from participants prior to vaccination and at 6 months post vaccination, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The lower detection limit for the assay was 0.08 micrograms/milliliter (µg/mL), and antibody levels below this limit were recorded as 0.04 µg/mL by the laboratory. Fold rises compare IgG antibody levels at the post-vaccination visit to that obtained just prior to vaccination. Participants are considered a responder if the antibody increase was four-fold or greater.
Time Frame: Prior to and 6 months following vaccination
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 279 | 287
participants | 264 | 1

9. Secondary Outcome: Number of Participants With a Four-Fold or Greater Rise in Serum IgG Antibody to Type III GBS at Month 8 Post-Vaccination
Description: Blood samples were collected from participants prior to vaccination and at 8 month post vaccination, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The lower detection limit for the assay was 0.08 micrograms/milliliter (µg/mL), and antibody levels below this limit were recorded as 0.04 µg/mL by the laboratory. Fold rises compare IgG antibody levels at the post-vaccination visit to that obtained just prior to vaccination. Participants are considered a responder if the antibody increase was four-fold or greater.
Time Frame: Prior to and 8 month following vaccination
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 275 | 278
participants | 256 | 1

10. Secondary Outcome: Number of Participants With a Four-Fold or Greater Rise in Serum IgG Antibody to Type III GBS at Month 10 Post-Vaccination
Description: Blood samples were collected from participants prior to vaccination and at 10 months post vaccination, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The lower detection limit for the assay was 0.08 micrograms/milliliter (µg/mL), and antibody levels below this limit were recorded as 0.04 µg/mL by the laboratory. Fold rises compare IgG antibody levels at the post-vaccination visit to that obtained just prior to vaccination. Participants are considered a responder if the antibody increase was four-fold or greater.
Time Frame: Prior to and 10 months following vaccination
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 271 | 262
participants | 250 | 1

11. Secondary Outcome: Number of Participants With a Four-Fold or Greater Rise in Serum IgG Antibody to Type III GBS at Month 12 Post-Vaccination
Description: Blood samples were collected from participants prior to vaccination and at 12 months post vaccination, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The lower detection limit for the assay was 0.08 micrograms/milliliter (µg/mL), and antibody levels below this limit were recorded as 0.04 µg/mL by the laboratory. Fold rises compare IgG antibody levels at the post-vaccination visit to that obtained just prior to vaccination. Participants are considered a responder if the antibody increase was four-fold or greater.
Time Frame: Prior to and 12 months following vaccination
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 271 | 274
participants | 245 | 2

12. Secondary Outcome: Number of Participants With a Four-Fold or Greater Rise in Serum IgG Antibody to Type III GBS at Month 14 Post-Vaccination
Description: Blood samples were collected from participants prior to vaccination and at 14 months post vaccination, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The lower detection limit for the assay was 0.08 micrograms/milliliter (µg/mL), and antibody levels below this limit were recorded as 0.04 µg/mL by the laboratory. Fold rises compare IgG antibody levels at the post-vaccination visit to that obtained just prior to vaccination. Participants are considered a responder if the antibody increase was four-fold or greater.
Time Frame: Prior to and 14 months following vaccination
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 258 | 261
participants | 231 | 3

13. Secondary Outcome: Number of Participants With a Four-Fold or Greater Rise in Serum IgG Antibody to Type III GBS at Month 16 Post-Vaccination
Description: Blood samples were collected from participants prior to vaccination and at 16 months post vaccination, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The lower detection limit for the assay was 0.08 micrograms/milliliter (µg/mL), and antibody levels below this limit were recorded as 0.04 µg/mL by the laboratory. Fold rises compare IgG antibody levels at the post-vaccination visit to that obtained just prior to vaccination. Participants are considered a responder if the antibody increase was four-fold or greater.
Time Frame: Prior to and 16 months following vaccination
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 256 | 260
participants | 228 | 2

14. Secondary Outcome: Number of Participants With a Four-Fold or Greater Rise in Serum IgG Antibody to Type III GBS at Month 18 Post-Vaccination
Description: Blood samples were collected from participants prior to vaccination and at 18 months post vaccination, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The lower detection limit for the assay was 0.08 micrograms/milliliter (µg/mL), and antibody levels below this limit were recorded as 0.04 µg/mL by the laboratory. Fold rises compare IgG antibody levels at the post-vaccination visit to that obtained just prior to vaccination. Participants are considered a responder if the antibody increase was four-fold or greater.
Time Frame: Prior to and 18 months following vaccination
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 264 | 261
participants | 229 | 1

15. Secondary Outcome: Number of Participants With a Serum IgG Antibody to Type III GBS Post-Vaccination of 5 µg/mL or Greater at Month 0
Description: Blood samples were collected from participants at each scheduled clinic visit beginning with Month 0 prior to vaccination, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The threshold for being considered seropositive was 5 µg/mL.
Time Frame: Month 0 prior to vaccination
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 325 | 325
participants | 25 | 18

16. Secondary Outcome: Number of Participants With a Serum IgG Antibody to Type III GBS Post-Vaccination of 5 µg/mL or Greater at Month 1 Post Vaccination
Description: Blood samples were collected from participants at each scheduled clinic visit and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The threshold for being considered seropositive was 5 µg/mL.
Time Frame: Month 1
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 304 | 303
participants | 192 | 12

17. Secondary Outcome: Number of Participants With a Serum IgG Antibody to Type III GBS Post-Vaccination of 5 µg/mL or Greater at Month 2 Post Vaccination
Description: as for outcome 16
Time Frame: Month 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 301 | 310
participants | 186 | 13

18. Secondary Outcome: Number of Participants With a Serum IgG Antibody to Type III GBS Post-Vaccination of 5 µg/mL or Greater at Month 4 Post Vaccination
Description: Blood samples were collected from participants at each scheduled clinic visit, and serum was assayed with an ELISA to measure IgG antibody levels to Type III GBS. The threshold for being considered seropositive was 5 µg/mL.
Time Frame: Month 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 289 | 298
participants | 174 | 12

19. Secondary Outcome: Number of Participants With a Serum IgG Antibody to Type III GBS Post-Vaccination of 5 µg/mL or Greater at Month 6 Post Vaccination
Description: as for outcome 18
Time Frame: Month 6
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 279 | 287
participants | 155 | 11

20. Secondary Outcome: Number of Participants With a Serum IgG Antibody to Type III GBS Post-Vaccination of 5 µg/mL or Greater at Month 8 Post Vaccination
Description: as for outcome 18
Time Frame: Month 8
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 275 | 278
participants | 151 | 9

21. Secondary Outcome: Number of Participants With a Serum IgG Antibody to Type III GBS Post-Vaccination of 5 µg/mL or Greater at Month 10 Post Vaccination
Description: as for outcome 18
Time Frame: Month 10
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 271 | 262
participants | 137 | 10

22. Secondary Outcome: Number of Participants With a Serum IgG Antibody to Type III GBS Post-Vaccination of 5 µg/mL or Greater at Month 12 Post Vaccination
Description: as for outcome 18
Time Frame: Month 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 271 | 274
participants | 136 | 10

23. Secondary Outcome: Number of Participants With a Serum IgG Antibody to Type III GBS Post-Vaccination of 5 µg/mL or Greater at Month 14 Post Vaccination
Description: as for outcome 18
Time Frame: Month 14
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 258 | 261
participants | 126 | 9

24. Secondary Outcome: Number of Participants With a Serum IgG Antibody to Type III GBS Post-Vaccination of 5 µg/mL or Greater at Month 16 Post Vaccination
Description: as for outcome 18
Time Frame: Month 16
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 256 | 260
participants | 122 | 8

25. Secondary Outcome: Number of Participants With a Serum IgG Antibody to Type III GBS Post-Vaccination of 5 µg/mL or Greater at Month 18 Post Vaccination
Description: as for outcome 18
Time Frame: Month 18
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 264 | 261
participants | 117 | 9

26. Secondary Outcome: Number of Participants Whose Vaginal Cultures Are Type III GBS Culture Negative Throughout the Study.
Description: Number of participants who were vaginal type III GBS negative was calculated throughout the the eighteen month post-vaccination follow-up period. Status at missed visits prior to loss to follow-up /final visit was imputed from the subsequent visit.
Time Frame: Every 2 months from time of vaccination up to 18 months post-vaccination.
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 325 | 325
Participants
  Always Vaginal Negative - False | 39 | 54
  Always Vaginal Negative - True | 286 | 271
Statistical Analysis 1: Comparison: GBS III-TT Vaccine vs Td Vaccine; A two-sided 5% level Fisher's exact test was used to test the null hypothesis of no difference in proportion of participants who were vaginal type III GBS negative throughout the study between treatment arms. The two-sided 5% Fisher's exact test was inverted to obtain a 95% confidence interval for the odds ratio; Test type: Superiority or Other; p = 0.120, Fisher Exact — The a priori threshold for statistical significance for the analysis of secondary endpoints was set at .05 without adjustment for multiplicity; Fisher's exact test was used to test no difference in proportions always vaginal GBS-III negative by arm to a two-sided alternative of a difference; Odds Ratio (OR) = 1.460, 95% CI 2-sided [0.917 to 2.34] — The OR was calculated from the 2x2 contingency table, and the 95% CI was obtained by inverting the 2-sided 5% level Fisher's exact, with GBS III-TT arm in the numerator and Td arm in the denominator so <1 favors the GBS III-TT arm

27. Secondary Outcome: Number of Participants Whose Vaginal Cultures Were Type III GBS Culture Positive.
Description: Number of participants whose vaginal swabs were type III GBS culture positive was calculated using data from the eighteen month post-vaccination follow-up period. Status at missed visits prior to loss to follow-up/final visit was imputed from the previous visit.
Time Frame: Every 2 months from time of vaccination up to 18 months post-vaccination.
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 325 | 325
Participants
  Month 1 - Missing | 5 | 2
  Month 1 - Negative | 313 | 314
  Month 1 - Positive | 7 | 9
  Month 2 - Missing | 8 | 7
  Month 2 - Negative | 303 | 310
  Month 2 - Positive | 14 | 8
  Month 4 - Missing | 24 | 15
  Month 4 - Negative | 292 | 301
  Month 4 - Positive | 9 | 9
  Month 6 - Missing | 25 | 22
  Month 6 - Negative | 293 | 291
  Month 6 - Positive | 7 | 12
  Month 8 - Missing | 34 | 29
  Month 8 - Negative | 282 | 279
  Month 8 - Positive | 9 | 17
  Month 10 - Missing | 41 | 38
  Month 10 - Negative | 279 | 273
  Month 10 - Positive | 5 | 14
  Month 12 - Missing | 48 | 42
  Month 12 - Negative | 272 | 266
  Month 12 - Positive | 5 | 17
  Month 14 - Missing | 52 | 51
  Month 14 - Negative | 268 | 259
  Month 14 - Positive | 5 | 15
  Month 16 - Missing | 58 | 56
  Month 16 - Negative | 260 | 257
  Month 16 - Positive | 7 | 12
  Month 18 - Missing | 61 | 62
  Month 18 - Negative | 256 | 255
  Month 18 - Positive | 7 | 8
  All Clinic Visits - Missing | 356 | 324
  All Clinic Visits - Negative | 3138 | 3126
  All Clinic Visits - Positive | 80 | 125
Statistical Analysis 1: Comparison: GBS III-TT Vaccine vs Td Vaccine; The proportion of vaginal swabs that were GBS III culture positive was estimated from a GEE model fit with binomial family, log-link, and exchangeable correlation. Point and robust interval estimates for vaccine efficacy, were obtained by transforming those for treatment effect in this model, and used to test the hypothesis of no efficacy; Test type: Superiority or Other; p = 0.089, Binomial regression, log-linear link — Significance was set at .05 without adjustment for multiplicity. Exchangeable correlation structure and GEE were used for repeated measures; The Wald test of treatment effect was used to test no difference in proportion of GBS III pos. by arm against a 2-sided alternative of a difference; Vaccine Efficacy, VE=1-RR=1-exp(ß) = 36, 95% CI [-7 to 61] — Estimate of vaccine efficacy and 95% CI were obtained by transforming the estimate of log relative risk for treatment effect and the robust Wald CI in the log-linear binomial regression model fit to the proportion of vaginal type III GBS swabs

28. Secondary Outcome: Number of Participants Whose Vaginal Cultures Were Persistently Type III GBS Culture Positive for Three or More Consecutive Visits
Description: Number of vaginal GBS III culture positive for 3+ consecutive visits was calculated from the post-vaccination visits over the 18 month follow-up. Status at missed visits prior to loss to follow-up/final visit was imputed from the subsequent visit.
Time Frame: Every 2 months from time of vaccination up to 18 months post-vaccination.
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 325 | 325
Participants
  Persistent Colonization - False | 318 | 312
  Persistent Colonization - True | 7 | 13
Statistical Analysis 1: Comparison: GBS III-TT Vaccine vs Td Vaccine; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; p = 0.256, Fisher Exact — [p-value comment as in outcome 26, analysis 1]; Fisher's exact test was used to test no difference in proportion persistently colonized by arm against a two-sided alternative of a difference; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.18 to 1.45] — The OR was calculated from the 2x2 contingency table, and the 95% CI was obtained by inverting the two-sided 5% level Fisher's exact test. The GBS III-TT arm is in the numerator and Td arm in the denominator, so a value <1 favors the GBS III-TT arm

29. Secondary Outcome: The Density of Type III GBS Cultured From Vaginal Swabs at Month 0
Description: The density of type III GBS is an ordinal response with six Density Levels: negative (lowest density, Score 0); broth only (Score 1); 1+ (Score 2); 2+ (Score 3); 3+ (Score 4); and 4+ (highest density, Score 5). The number of swabs with each score was tabulated from swabs collected at Month 0 prior to vaccination.
Time Frame: Month 0
Population: as for outcome 2
Measure: Number; unit: Swabs
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 325 | 325
Swabs
  Negative | 321 | 320
  Broth only | 0 | 1
  1+ | 0 | 0
  2+ | 0 | 0
  3+ | 0 | 0
  4+ | 4 | 4

30. Secondary Outcome: The Density of Type III GBS Cultured From Vaginal Swabs at Month 1
Description: The density of type III GBS is an ordinal response with six Density Levels: negative (lowest density, Score 0); broth only (Score 1); 1+ (Score 2); 2+ (Score 3); 3+ (Score 4); and 4+ (highest density, Score 5). The number of swabs with each score was tabulated from swabs collected at Month 1. Density at missed visits prior to loss to follow-up/final visit was imputed from the subsequent visit.
Time Frame: Month 1
Population: as for outcome 2
Measure: Number; unit: Swabs
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 323 | 320
Swabs
  Negative | 314 | 313
  Broth only | 1 | 1
  1+ | 0 | 1
  2+ | 1 | 1
  3+ | 2 | 3
  4+ | 5 | 1

31. Secondary Outcome: The Density of Type III GBS Cultured From Vaginal Swabs at Month 2
Description: The density of type III GBS is an ordinal response with six Density Levels: negative (lowest density, Score 0); broth only (Score 1); 1+ (Score 2); 2+ (Score 3); 3+ (Score 4); and 4+ (highest density, Score 5). The number of swabs with each score was tabulated from swabs collected at Month 2. Density at missed visits prior to loss to follow-up/final visit was imputed from the subsequent visit.
Time Frame: Month 2
Population: as for outcome 2
Measure: Number; unit: Swabs
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 318 | 317
Swabs
  Negative | 310 | 303
  Broth only | 0 | 1
  1+ | 0 | 1
  2+ | 2 | 1
  3+ | 1 | 2
  4+ | 5 | 9

32. Secondary Outcome: The Density of Type III GBS Cultured From Vaginal Swabs at Month 4
Description: The density of type III GBS is an ordinal response with six Density Levels: negative (lowest density, Score 0); broth only (Score 1); 1+ (Score 2); 2+ (Score 3); 3+ (Score 4); and 4+ (highest density, Score 5). The number of swabs with each score was tabulated from swabs collected at Month 4. Density at missed visits prior to loss to follow-up/final visit was imputed from the subsequent visit.
Time Frame: Month 4
Population: as for outcome 2
Measure: Number; unit: Swabs
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 310 | 301
Swabs
  Negative | 301 | 292
  Broth only | 2 | 0
  1+ | 1 | 2
  2+ | 2 | 0
  3+ | 1 | 3
  4+ | 3 | 4

33. Secondary Outcome: The Density of Type III GBS Cultured From Vaginal Swabs at Month 6
Description: The density of type III GBS is an ordinal response with six Density Levels: negative (lowest density, Score 0); broth only (Score 1); 1+ (Score 2); 2+ (Score 3); 3+ (Score 4); and 4+ (highest density, Score 5). The number of swabs with each score was tabulated from swabs collected at Month 6. Density at missed visits prior to loss to follow-up/final visit was imputed from the subsequent visit.
Time Frame: Month 6
Population: as for outcome 2
Measure: Number; unit: Swabs
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 303 | 300
Swabs
  Negative | 291 | 293
  Broth only | 1 | 2
  1+ | 0 | 0
  2+ | 1 | 0
  3+ | 2 | 2
  4+ | 8 | 3

34. Secondary Outcome: The Density of Type III GBS Cultured From Vaginal Swabs at Month 8
Description: The density of type III GBS is an ordinal response with six Density Levels: negative (lowest density, Score 0); broth only (Score 1); 1+ (Score 2); 2+ (Score 3); 3+ (Score 4); and 4+ (highest density, Score 5). The number of swabs with each score was tabulated from swabs collected at Month 8. Density at missed visits prior to loss to follow-up/final visit was imputed from the subsequent visit.
Time Frame: Month 8
Population: as for outcome 2
Measure: Number; unit: Swabs
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 296 | 291
Swabs
  Negative | 279 | 282
  Broth only | 3 | 1
  1+ | 0 | 0
  2+ | 0 | 2
  3+ | 1 | 2
  4+ | 13 | 4

35. Secondary Outcome: The Density of Type III GBS Cultured From Vaginal Swabs at Month 10
Description: The density of type III GBS is an ordinal response with six Density Levels: negative (lowest density, Score 0); broth only (Score 1); 1+ (Score 2); 2+ (Score 3); 3+ (Score 4); and 4+ (highest density, Score 5). The number of swabs with each score was tabulated from swabs collected at Month 10. Density at missed visits prior to loss to follow-up/final visit was imputed from the subsequent visit.
Time Frame: Month 10
Population: as for outcome 2
Measure: Number; unit: Swabs
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 287 | 284
Swabs
  Negative | 273 | 279
  Broth only | 2 | 1
  1+ | 0 | 0
  2+ | 3 | 1
  3+ | 3 | 0
  4+ | 6 | 3

36. Secondary Outcome: The Density of Type III GBS Cultured From Vaginal Swabs at Month 12
Description: The density of type III GBS is an ordinal response with six Density Levels: negative (lowest density, Score 0); broth only (Score 1); 1+ (Score 2); 2+ (Score 3); 3+ (Score 4); and 4+ (highest density, Score 5). The number of swabs with each score was tabulated from swabs collected at Month 12. Density at missed visits prior to loss to follow-up/final visit was imputed from the subsequent visit.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number; unit: Swabs
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 283 | 277
Swabs
  Negative | 266 | 272
  Broth only | 2 | 0
  1+ | 0 | 0
  2+ | 3 | 1
  3+ | 1 | 2
  4+ | 11 | 2

37. Secondary Outcome: The Density of Type III GBS Cultured From Vaginal Swabs at Month 14
Description: The density of type III GBS is an ordinal response with six Density Levels: negative (lowest density, Score 0); broth only (Score 1); 1+ (Score 2); 2+ (Score 3); 3+ (Score 4); and 4+ (highest density, Score 5). The number of swabs with each score was tabulated from swabs collected at Month 14. Density at missed visits prior to loss to follow-up/final visit was imputed from the subsequent visit.
Time Frame: Month 14
Population: as for outcome 2
Measure: Number; unit: Swabs
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 274 | 273
Swabs
  Negative | 259 | 268
  Broth only | 3 | 0
  1+ | 2 | 1
  2+ | 1 | 0
  3+ | 4 | 2
  4+ | 5 | 2

38. Secondary Outcome: The Density of Type III GBS Cultured From Vaginal Swabs at Month 16
Description: The density of type III GBS is an ordinal response with six Density Levels: negative (lowest density, Score 0); broth only (Score 1); 1+ (Score 2); 2+ (Score 3); 3+ (Score 4); and 4+ (highest density, Score 5). The number of swabs with each score was tabulated from swabs collected at Month 16. Density at missed visits prior to loss to follow-up/final visit was imputed from the subsequent visit.
Time Frame: Month 16
Population: as for outcome 2
Measure: Number; unit: Swabs
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 269 | 267
Swabs
  Negative | 257 | 260
  Broth only | 2 | 2
  1+ | 1 | 1
  2+ | 1 | 0
  3+ | 3 | 0
  4+ | 5 | 4

39. Secondary Outcome: The Density of Type III GBS Cultured From Vaginal Swabs at Month 18
Description: The density of type III GBS is an ordinal response with six Density Levels: negative (lowest density, Score 0); broth only (Score 1); 1+ (Score 2); 2+ (Score 3); 3+ (Score 4); and 4+ (highest density, Score 5). The number of swabs with each score was tabulated from swabs collected at Month 18. Density at missed visits prior to loss to follow-up/final visit was imputed from the subsequent visit.
Time Frame: Month 18
Population: as for outcome 2
Measure: Number; unit: Swabs
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Number analyzed (Participants) | 263 | 263
Swabs
  Negative | 255 | 256
  Broth only | 0 | 2
  1+ | 1 | 0
  2+ | 1 | 1
  3+ | 2 | 0
  4+ | 4 | 4

ADVERSE EVENTS:
Time Frame: Solicited reactogenicity was collected for 7 days after vaccination. Unsolicited serious and non-serious adverse events were collected throughout the 18-month duration of subject participation.
Description: The Safety Analysis Cohort is comprised of all vaccinated women, categorized according to the product received, regardless of their randomized assignment. Due to vaccination errors, the number of participants in the Td group for the Safety Analysis Cohort (n=337) exceeds the number randomized to this group (n=334).
Groups:
- GBS III-TT Vaccine: The experimental arm received a single dose of GBS III-TT vaccine administered intramuscularly (IM) containing 50 mcg of GBS III capsular polysaccharide and 32 mcg of tetanus toxoid. The Safety Analysis Cohort is comprised of all vaccinated women, categorized according to the product received, regardless of their randomized assignment.
- Td Vaccine: The control group received a single dose of tetanus and diptheria toxoids adsorbed for adult use (Td vaccine). The Safety Analysis Cohort is comprised of all vaccinated women, categorized according to the product received, regardless of their randomized assignment.
Arm/Group | GBS III-TT Vaccine | Td Vaccine
Serious Adverse Events (participants affected / at risk) | 14/326 | 22/337
Other Adverse Events (participants affected / at risk) | 304/326 | 320/337
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBS III-TT Vaccine (N=326) | Td Vaccine (N=337)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Polytraumatism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Psychiatric disorders) | 0 (0) | 1 (1)
Throat lesion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBS III-TT Vaccine (N=326) | Td Vaccine (N=337)
Nasopharyngitis (Infections and infestations) | 56 (61) | 55 (71)
Vaginitis bacterial (Infections and infestations) | 44 (51) | 61 (90)
Fungal infection (Infections and infestations) | 44 (52) | 45 (68)
Headache (Nervous system disorders) | 35 (37) | 44 (52)
Urinary tract infection (Infections and infestations) | 35 (46) | 29 (34)
Sinusitis (Infections and infestations) | 23 (33) | 30 (38)
Vulvovaginal mycotic infection (Infections and infestations) | 18 (19) | 19 (26)
Influenza (Infections and infestations) | 14 (15) | 19 (21)
Tenderness (General disorders) | 234 (234) | 276 (276)
Pain (at Injection Site) (General disorders) | 175 (175) | 223 (223)
Headache (Nervous system disorders) | 130 (130) | 119 (119)
Malaise (General disorders) | 103 (103) | 111 (111)
Myalgia (Musculoskeletal and connective tissue disorders) | 91 (91) | 112 (112)
Nausea (Gastrointestinal disorders) | 54 (54) | 61 (61)
Injection site swelling (General disorders) | 32 (32) | 54 (54)
Injection site erythema (General disorders) | 39 (39) | 45 (45)
Pyrexia (General disorders) | 33 (33) | 32 (32)
Chills (General disorders) | 30 (30) | 33 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less